CLINICAL TRIAL: NCT04826341
Title: A Phase I/II Study of Sacituzumab Govitecan Plus Berzosertib in Small Cell Lung Cancer, Extra-Pulmonary Small Cell Neuroendocrine Cancer and Homologous Recombination-Deficient Cancers Resistant to PARP Inhibitors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000144; 000144-C
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-10

CONDITIONS: HRD Cancer; SCLC; Advanced Solid Tumors
Keywords: PARPi resistance; ATR inhibition; targeted DNA-damaging chemotherapy; Antibody-Drug Conjugate; topoisomerase-I inhibiting camptothecin
MeSH Terms: interventions — berzosertib; sacituzumab govitecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I (Experimental): Dose escalated Sacituzumab Govitecan and Berzosertib
  Interventions: Drug: Berzosertib; Drug: Sacituzumab Govitecan
- 2/Phase II (Experimental): Sacituzumab Govitecan and Berzosertib treatment with identified MTD based on phase I.
  Interventions: Drug: Berzosertib; Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Berzosertib — Berzosertib will be supplied as 20 mg/mL M6620 to be diluted with 5% dextrose in water solution before intravenous infusion.
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan will be administered as an intravenous infusion once weekly on Days 1 and 8 of 21-day treatment cycles.

SUMMARY:
Background:

Small cell lung cancer and PARP inhibitor resistant tumors are aggressive cancers. Current treatments for people with these tumors yield little benefit. Researchers want to see if a combination of drugs can help.

Objective:

To find a safe combination of sacituzumab govitecan and berzosertib and to see if this will cause small cell lung cancer and PARP inhibitor resistant tumors to shrink.

Eligibility:

People ages 18 and older with a solid tumor, small cell lung cancer, or a homologous recombination-deficient cancer that is resistant to PARP inhibitors

Design:

Participants will be screened with:

Standard clinical exams and tests

EKG to test the heart

Medical documentation to confirm cancer diagnosis

Participants will get sacituzumab govitecan by vein on days 1 and 8 of each 21-day cycle. They will get berzosertib by vein on days 2 and 9. Treatment will continue as long as they can tolerate the drugs and their tumors are either stable or getting better.

Before treatment and at least once per cycle, participants will have a physical exam and blood tests. Before treatment and every 2 or 3 cycles, they will have a CT scan. They will have a contrast agent injected into a vein for the scan.

Participants will give blood and hair samples and tumor biopsies for research. Biopsies will be taken with a small needle under imaging guidance.

After they stop treatment, participants will have a visit 1 month later. They will then be contacted by phone or email every 3 months for the rest of their lives.

DETAILED DESCRIPTION:
Background:

Several small molecule poly-(ADP)-ribose polymerase inhibitors (PARPi) have been approved by the FDA for multiple cancers with homologous recombination (HR) deficiencies. Despite their measurable initial benefit, PARPi resistance is a major problem in the clinic. There are no established standards for care of patients who have disease progression after PARPi.

Small cell lung cancer (SCLC) is an aggressive cancer with poor prognosis. Despite being chemo-sensitive initially, the tumors are invariably chemo-resistant at recurrence. Currently available therapies for patients who have disease progression after chemotherapy yield limited benefit, and most patients die within months of relapse.

Extra pulmonary small cell neuroendocrine (EP-SCNC) cancers are exceedingly rare cancers with small cell morphology arising from non-lung primary sites. The striking responses that we see to combinations of TOP1 and ATR inhibitors suggest high replication stress in these tumors, and provide compelling rationale to rigorously investigate the effect of this combination using a less toxic combination of IMMU132 and berzosertib.

In preclinical studies, ataxia telangiectasia and Rad3-related protein (ATR) inhibition can overcome PARPi/chemotherapy-resistance in tumors with restored HR or restored fork protection. However, combinations of DNA damage response inhibitors and chemotherapy may be challenging in clinic due to overlapping toxicities, specifically myelosuppression.

To mitigate some of the overlapping toxicities relating to myelosuppression, we have proposed a strategy that incorporates tumor targeted DNA-damaging chemotherapy delivery (using approaches such as antibody drug conjugates) and dose scheduling of ATR inhibitors.

Sacituzumab govitecan is an antibody-drug conjugate, comprising a topoisomerase-I inhibiting camptothecin, SN-38, linked to a humanized antibody targeting trophoblastic cell-surface antigen 2 (Trop-2), and is FDA approved as Trodelvy (Trademark) for triple-negative breast cancer patients and hormone receptor-positive, HER2-negative breast cancer.

Berzosertib is a potent and selective kinase inhibitor of ATR in phase I and II clinical trials as a single agent and in combination with chemotherapy, radiation and other anticancer agents.

We hypothesize that a combination of berzosertib with sacituzumab govitecan will provide an effective therapeutic option for patients with PARPi resistant tumors and chemotherapy-resistant SCLCs. This combination will also be evaluated for efficacy in EP-SCNC and HRD positive tumors.

Primary objectives:

Phase I: To identify the maximum tolerated dose (MTD) of sacituzumab govitecan in combination with berzosertib.

Phase II HRD cohort: To assess the efficacy with respect to objective response rate (ORR) of the combination of sacituzumab govitecan and berzosertib in previously treated participants with HRD.

Phase II SCLC cohort: To assess the efficacy with respect to ORR of the combination of sacituzumab govitecan and berzosertib in previously treated participants with SCLC.

Eligibility:

All phases: Subjects must be >= 18 years of age and have a performance status (ECOG) <= 2.

Phase I: Adult participants with advanced solid tumors with progression on at least one prior chemotherapy.

Phase II HRD cohort: Known HRD cancer and documented evidence of germline or somatic BRCA mutation or other HRD germline mutation, or tumor is HRD positive; progressive disease while taking a PARPi as a previous therapy or within 6 months of completing PARPi therapy.

Phase II SCLC or EP-SCNC cohort: Recurrent SCLC or EP-SCNC after at least one prior platinum-based therapy.

Design:

This is a Phase I/II, open label clinical trial identifying the maximum tolerated dose (MTD) of sacituzumab govitecan in combination with berzosertib in a phase I trial, and assessing the efficacy with respect to clinical response rate of a combination of sacituzumab govitecan and berzosertib as treatment of subjects with recurrent SCLC, EPSCNC and HRD positive tumors. The accrual ceiling will be set to 120 for this study.

Participants will receive sacituzumab govitecan on days 1 and 8 and berzosertib on days 2 and 9, administered every 21 days (1 cycle), until disease progression or development of intolerable side effects.

Blood, hair follicles, and tumor will be collected at various time points to support the exploratory objectives.

The Phase I will follow a 3+3 design: dose will be escalated in cohorts of 3-6 participants each with the individual dose of berzosertib and sacituzumab govitecan increased in successive dose levels.

The phase II HRD cohort and phase II SCLC cohort will be conducted using a Simon two-stage Minimax design in order to rule out an unacceptably low 5% response rate (p0=0.05) for HRD and 10% (p=0.10) response rate for SCLC in favor of a targeted response rate of 20% (p1=0.20) and 30% (p1=0.30), respectively.

A small cohort of extra-pulmonary small cell neuroendocrine cancers (EP-SCNC) will also be included to provide limited assessment of efficacy in this rare population.

ELIGIBILITY:
* INCLUSION CRITERIA:

All phases and cohorts

-Subjects must not have received chemotherapy or undergone major surgery within 2 weeks and radiotherapy within 24 hours prior to cycle 1 day 1.

* Age >=18 years. Because no dosing or adverse event data are currently available on the use of sacituzumab govitecan in combination with and berzosertib in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status <=2
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >=3,000/mcL
  * Hemoglobin >=9.0g/dL
  * absolute neutrophil count >=1,500/mcL
  * platelets >=100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits

OR

--creatinine clearance >=30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal

(calculated by Cockcroft-Gault formula).

* Participants with neurologically stable brain metastases defined as asymptomatic metastasis, or treated metastasis having no evidence of progression or hemorrhage for at least 2 weeks after treatment (including brain radiotherapy) may be included. Participants must be off any systemic corticosteroids for the treatment of brain metastases for at least 7 days prior to enrollment.
* Participants with previously treated with topoisomerase 1/2 inhibitors can be enrolled.
* The effects of the combined study drugs on the developing human fetus are unknown. For this reason and because study agents as well as other therapeutic agents used in this trial are known to be teratogenic, individuals of child-bearing potential and individuals who can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, while taking the study drugs and for 6 months after the administered study drug (berzosertib or sacituzumab govitecan).
* Ability of subject to understand and the willingness to sign a written informed consent document.

Phase I

-Participants with histologically or cytologically confirmed advanced solid tumors with progression on at least one prior chemotherapy.

Phase II HRD cohort

-Known HRD cancer and documented evidence of at least ONE or MORE of the following:

--Pathogenic or likely pathogenic somatic mutation or inactivating alteration of a gene involved in homologous recombination (BRCA1, BRCA2, ATM, BRIP1, BARD1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, or RAD54L) repair in the tumor. Local testing in Clinical Laboratory Improvement Act (CLIA)-certified laboratory will be accepted. No

variants of uncertain significance (VUS) will be allowed.

* If this alteration is identified in a circulating tumor deoxyribonucleic acid (ctDNA) assay, the variant-allele fraction must be > 20% to indicate relevance to predominant tumor clone
* Mutation in one or more other genes involved in homologous DNA recombination repair in the tumor may be included at investigator's

discretion

---Homologous recombination repair deficiency by genomic signature in the tumor by BROCA-HR, Foundation One or equivalent assay

--Presence of pathogenic or likely pathogenic germline mutation/variant in BRCA1, BRCA2, ATM, BRIP1, BARD1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, or RAD54L. Germline mutations in other HR genes will be considered at investigator's discretion. Local testing in Clinical Laboratory Improvement Act (CLIA)-certified laboratory will be accepted. No variants of uncertain significance (VUS) will be allowed.

* Participants must have measurable disease, per RECIST 1.1.
* Participants must have at least one lesion deemed safe to biopsy and be willing to undergo mandatory biopsies (Pre-treatment, On-Treatment, PD). Up to 10 participants with non-biopsiable disease may be enrolled.
* Participants should have demonstrated progressive disease while taking a PARPi as a previous therapy or within 6 months of completing PARPi therapy. Response to prior PARPi is not required.
* Participants may have received chemotherapy in the interval between PARPi and enrollment.

Phase II SCLC and EP-SCNC

* Recurrent histologically or cytologically confirmed SCLC or EP-SCNC after at least one prior platinum-based therapy.
* Participants must have measurable disease, per RECIST 1.1.
* Participants must have at least one lesion deemed safe to biopsy and be willing to undergo mandatory biopsies (Pre-Treatment, On-Treatment, PD). Up to 10 participants with non-biopsiable disease may be enrolled.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents or concurrent systemic anti-cancer therapies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs or other agents used in study.
* Participants with symptomatic brain metastasis.
* Participants who require treatment with strong inhibitors or inducers of CYP3A or with UGT1A1 inhibitors during the planned period of investigational treatment with sacituzumab govitecan.
* Participants known to be homozygous for the UGT1A1*28 variant allele with severely reduced UGT1A1 activity.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant individuals are excluded from this study because study drugs have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study drugs, breastfeeding should be discontinued if the mother is treated with the study drugs. These potential risks may also apply to other agents used in this study.
* Participants with myelosuppressive disorders or acute myeloid leukemia.
* HIV positive participants with the following exception: Patients with long-standing (>5 years) HIV on antiretroviral therapy > 1 month (undetectable HIV viral load and CD4 count > 150 cells/microL) may be eligible if the principal investigator determines no anticipated clinically significant drug-drug interactions.
* Participants with evidence of chronic hepatitis B virus (HBV) infection, unless the HBV viral load is undetectable and participant is on suppressive therapy, if indicated.
* HCV infected participants with the following exceptions: Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase II: ORR | Disease progression
  In phase II, in each cohort, the fraction of participants who experience a PR or CR will be reported along with a 95% confidence interval.
Phase I: MTD | Phase I
  In phase I, the toxicities identified at each dose level will be reported, by dose level, type, and grade.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Disease progression
  Progression free survival (PFS) will be calculated from on-study date until date of progression or death without progression, using the Kaplan-Meier method accompanied by determination of the median and its 95% confidence interval.
Overall survival (OS) | Death
  Overall survival (OS) will be calculated from the on-study date until date of death.
Toxicity grade and type | during treatment
  To assess safety and tolerability in phase II cohort in PARP inhibitor-resistant HRD tumors and previously treated SCLC, the toxicity grade and type will be reported for all patients treated on the two cohorts.
Duration of response | Disease progression
  Duration of response will be calculated by the Kaplan-Meier method (accompanied by determination of the median and its 95% confidence interval), starting at date response was identified until progression or the response is declared to have ended, if the participants have a PR or CR.
Safety and tolerability | during treatment
  Safety and tolerability of the combination will be reported by describing Adverse Events (AE) per CTCAE v5.0, by dose level, and type and grade of toxicity. This will be focused on phase I but also reported in phase II.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000144-C.html